CLINICAL TRIAL: NCT04693169
Title: [Al18F]PSMA137 PET/CT Imaging for PSMA-Positive Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Hua Zhu, Associate Professor, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020KT154
Record Dates: First submitted 2020-12-30; First posted 2021-01-05 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Prostate Cancer
Keywords: PSMA
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [Al18F]PSMA137 PET/CT imaging (Experimental): All study participants will be allocated to this arm (single-arm study).Study participants will undergo [Al18F]PSMA137 PET/CT scans.
  Interventions: Drug: 11C-Choline

INTERVENTIONS:
Drug: 11C-Choline — 1、PSMA137 labeled with [Al18F] will be used as a molecular imaging tracer for PET/CT scanning。 2、11C-choline (0.05-0.1mCi/kg) was injected intravenously in a week after the [Al18F]PSMA137 PET/CT examination, and imaging of the head and body cadres was performed 20 min after the injection using Philips Gemini TF16 or Siemens Biograph M-CT flow PET/CT
  Other Names: 11C-CH

SUMMARY:
To investigate the radioactive uptake of [Al 18 F]PSMA137 in PCa patients, and evaluate the ability of [Al 18 F]PSMA137 to detect PSMA overexpression in PCa patients (especially those with recurrent or advanced PCa).To provide an approach for screening patients high expression of PSMA, efficacy monitoring, drug resistance and early warning of recurrence and metastasis to achieve the individualized antitumor treatment of targeted drugs.

DETAILED DESCRIPTION:
Prostate cancer (PCa) is the most common malignant tumor in the male reproductive system, and its prognosis and treatment mainly depend on the discovery of the primary disease and the early stage of metastasis, while traditional imaging and histological methods are difficult to meet the clinical requirements for the early diagnosis and accurate staging of PCa.Positron emission tomography (PET) has the characteristics of precision and non-invasive, so the development of PCa targeted molecular probe is of great significance for improving the specificity and accuracy of PCa diagnosis.

PSMA is a highly specific prostatic epithelial membrane antigen, which is highly expressed in solid tumors such as Prostate cancer. More than 90% of Prostate cancer cells express PSMA, so PSMA can be used as an important imaging target for Prostate cancer.

The radionuclides used for PET imaging include 18F (T 1/2 =109.8min), which has a suitable half-life and cyclotron preparation to enable the high yield synthesis of 18F labeled tracer, so it can be used in more patients and provided to other departments without on-site tracer production facilities.In addition, coordination labeling method is simple, easy to realize automatic synthesis technology and medicine box preparation.Therefore, 18F-labeled PSMA targeted molecular probe is a hot spot in the diagnosis of prostate cancer.

[Al18F]PSMA137 is a novel PSMA targeted tracer labeled with 18F. NOTA is used as a bifunctional chelating agent to facilitate better chelation with Al18F. It has a higher tumor uptake and a faster metabolism in normal organs with a lower background.[Al18F]PSMA137, as a novel targeted molecular probe, shows excellent properties in tumor cell uptake.This project provides research on [Al18F]PSMA137 PET/CT imaging for patients with suspected PCa, and provides basis for early diagnosis of PCa, formulation of treatment plan and efficacy evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Men over 18 years of age need to undergo [Al18F]PSMA137 PET/CT examination for suspected prostate cancer.
* The patients can fully understand and voluntarily participate in this experiment, and sign the informed consent.

Exclusion Criteria:

* Significant hepatic or renal dysfunction;
* Patients with malignant tumors other than prostate cancer within 2 years;
* Ready to pregnant;
* The patient can not tolerate all clinical tests.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-01-15 (Actual); Primary Completion 2024-06-12 (Estimated); Study Completion 2024-12-12 (Estimated)

PRIMARY OUTCOMES:
SUV（standardized uptake value） | 2 years
  SUV is a semi-quantitative analysis index to describe the radioactive uptake of lesions, which has certain reference value for differentiating benign and malignant lesions。 The uptake of the tracer （[Al18F]PSMA137） in the primary and metastatic tumor lesions by measuring SUV on PET/CT

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No